CLINICAL TRIAL: NCT04131374
Title: Going Down Memory Lane: Developing a Technological Intervention for Older Adults Living With Dementia and Their Family Caregivers
Brief Title: Going Down Memory Lane: A Technological Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: The Brenda Strafford Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB18-1902
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Dementia
Keywords: Caregivers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: We will select 5 people living with dementia and their family caregiver. All participants will participate in developing their own tailored VR scenario and receive a weekly VR intervention (30 minutes) over a period of 10 weeks.
  Participants (i.e. person living with dementia, family caregiver) will complete outcome measures at baseline (week 1), mid-intervention (week 5), the conclusion of intervention (week 10), and 5-weeks following the intervention (week 15).
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Intervention (Experimental): Virtual Reality Intervention: Each Person Living with Dementia-caregiver dyad will receive 10 weekly sessions of tailored reminiscence therapy delivered via virtual reality. Each session will last for a period of 15-30 minutes.
  Interventions: Behavioral: Reminiscence Therapy

INTERVENTIONS:
Behavioral: Reminiscence Therapy — Virtual reality scenarios will be used to delivered reminiscence therapy with each caregiving dyad (i.e. person living with dementia; family member).

SUMMARY:
Over 90% of people living with dementia (PLWD) experience behavioural and psychological symptoms of dementia, including apathy, depression, sleep disruptions, wandering, repetitive behaviours and anxiety. These symptoms can result in poor quality of life, burden for caregivers, and an increased risk for physical abuse of PLWD.

This study aims to evaluate the acceptability, feasibility, and efficacy of a reminiscence therapy intervention using virtual reality technology, to reduce symptoms associated with dementia in older adults. Further, the investigators will assess if the intervention improved the quality of life of participants and the relationship between the person living with dementia and their caregiver.

DETAILED DESCRIPTION:
Background: Over 90% of people living with dementia (PLWD) experience behavioural and psychological symptoms of dementia (BPSD) including apathy, depression, sleep disruptions, wandering, repetitive behaviours and anxiety. BPSD can also result in poor quality of life, burden for caregivers, and an increased risk for physical abuse of PLWD. Incorporating the family caregiver into the plan of care may improve satisfaction and lower the burden associated with providing care for PLWD in a nursing home. New evidence suggests limited benefits of pharmacological interventions and increased risks for adverse events for PLWD. Results from systematic reviews suggest that Reminiscence Therapy (RT) has positive outcomes for people with dementia, such as elevated mood, improved cognition and enhanced behaviours. An additional systematic review indicates there are significant benefits of using information communication technology (ICT) for RT interventions. Virtual reality (VR) is emerging as a promising non-pharmacological approach for reducing symptoms of dementia and allows for tailoring of technological intervention to the user. To our knowledge, VR scenarios have never been developed as a RT intervention for PLWD and their caregiver.

Purpose and Objectives: The purpose of this innovative, interdisciplinary study is to design and test a VR technological intervention with older adults with dementia and their caregivers, guided by RT. The main research question is: Can a tailored VR intervention reduce BPSD among PLWD and improve the caregiving relationship? Study objectives are to: (1) interview caregiving dyads to collect historical data to create tailored VR interventions using iterative design process; (2) test VR intervention with the caregiving dyads to assess: (a) impact on BPSD among PLWD and quality of the relationship between the PLWD and their family caregiver; and (b) impact of the intervention on family caregiver outcomes.

Study Design: The proposed feasibility (repeated measure design) study will be conducted in two phases and will include qualitative and quantitative data collection.

In PHASE 1 (design), 5 PLWD and their family caregiver will participate in 2-3 interviews which will be used to generate their personalized VR scenarios.

In PHASE 2 (testing), the tailored VR sessions from phase 1, will be used as a weekly intervention with each caregiving dyad over 10 weeks. Each tailored session will be 30 minutes in length. Participants will be positioned beside each other in stabilizing chairs, both wearing the 3D glasses, and viewing the same scenario.

Participants will be evaluated at 4-time points [week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5-week follow up)]. Using previously validated measures, participants living with dementia will be assessed on:

1. Behavioural or psychological symptom of dementia (Neuropsychiatric Inventory- Questionnaire)
2. Perceptions of person-centred care (Person-centered Climate Questionnaire-patient version)
3. Quality of Life (World Health Organization Quality of Life Instrument)

Family Caregiving participants will be assessed on:

1. Caregiving experience (A. Caregiver Reaction Scale, and B. Modified Caregiver Strain Index)
2. Quality of Life (World Health Organization Quality of Life Instrument)

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with moderate stages (stages 1-3) of dementia
* able to speak and read English
* caregivers should be a family caregiver of the person living with dementia
* caregivers should be 18 years of age or older
* caregivers should be able to speak and read English

Exclusion Criteria:

* physical limitations that prevent the application of research instruments (i.e. Virtual Reality technology)
* caregivers that do no reside in the same city as the person living with dementia, which prevents them from attending the weekly sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in participant's Behavioral or Psychological symptoms of dementia | week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5 week follow up)
  Caregivers will complete the Neuropsychiatric Inventory-Questionnaire (NPI-Q). This is a self-administered scale that is completed by the family caregiver. The scale has 12 items (dichotomous response) related to the behavioral or psychological symptoms of dementia. If the respondent indicates 'Yes,' a symptom is present, they are asked to rate the severity and distress. The severity of the symptoms is rated on a 3 point scale (mild, moderate, severe) over the last three months, and Distress is measured on a 5 point scale (no distress, minimal, mild, moderate, severe, very severe) indicating the amount of distress on the caregiver. The individual items are added together for an overall Severity and Distress score (minimum score 0- maximum score 96). Higher scores reflect worsening behavioural/psychological symptoms of dementia and increased caregiver distress.

SECONDARY OUTCOMES:
Change from baseline in participant's perception of person-centred care | week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5 week follow up)
  Participants living with dementia will complete the Person-Centered Climate Questionnaire (patient version). The Person-Centered Climate Questionnaire (patient version) measures the extent to which the psychosocial environment of a setting is perceived as being person-centred. The tool has 17 items in which respondents are asked to agree or disagree by selecting an answer on a 6 point scale, from "No, I disagree completely" to "Yes, I agree completely." The items are added together for an overall score, with a minimum scale score of 0 and a maximum scale score of 85. Higher scores reflect a more person-centred environment.
Change from baseline in the participant's quality of life | week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5 week follow up)
  Participants living with dementia will complete the World Health Organization Quality of Life Instrument (Brief). The World Health Organization Quality of Life Brief Instrument measures the quality of life through the following four domains and two overall health and quality of life items: physical health, psychological, social relationships, and environment. The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life. There are three items that are reversed scored. The possible raw score ranges for each domain are as follows: Physical Health =28, Psychological =24, Social Relationships =12, and environment =32.
Change from baseline in the caregiver's quality of life | week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5 week follow up)
  Caregivers will complete the World Health Organization Quality of Life Instrument (Brief). The World Health Organization Quality of Life Brief Instrument measures the quality of life through the following four domains and two overall health and quality of life items: physical health, psychological, social relationships, and environment. The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life. There are three items that are reversed scored. The possible raw score ranges for each domain are as follows: Physical Health =28, Psychological =24, Social Relationships =12, and environment =32.
Change from baseline in the caregiver's experience in caregiving | week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5 week follow up)
  Caregivers will complete the Caregiver Reaction Scale. The Caregiver Reaction Scale is a brief self-report measure, containing 8 subscales related to multiple dimensions of caregiving: caregiver's role captivity, overload, relational deprivation, caregiving competence, personal gain, family beliefs and actions and employment. The scale has a total of 54 items, which are scored on a 4-point scale where 1=not at all and 4 = completely. Scores for each subscale are averaged, with higher mean scores indicated high levels of negative and positive experiences. Subscales scores are interpreted independently.
Change from baseline in the caregiver's experience of caregiver strain | week 1 (baseline), week 5 (mid-intervention), week 10 (conclusion of intervention) and week 15 (5 week follow up)
  Caregivers will complete the Modified Caregiver Strain Index. The tool has 13 items that measure strain related to care provision, and it measures the following domains: financial, physical, psychological, social, and personal. Each item is scored on a 3 point scale (yes [2 points], sometimes [1 point], no [0 points'). Scores range from 0 to 26, and a higher score indicated a higher level of caregiver strain.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Duffett-Leger, PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No